CLINICAL TRIAL: NCT06114420
Title: Surgical Treatment and Molecular Marker Exploration of Locally Recurrent Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, ZHENGZHAOXU, M.D., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: CancerIHCAMS-NCC4237
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Locally Recurrent Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with local recurrence
  Interventions: Procedure: salvage surgery
- patients without local recurrence

INTERVENTIONS:
Procedure: salvage surgery — Some patients who cannot undergo surgery
  Other Names: adjuvant treatment
  Groups: patients with local recurrence

SUMMARY:
This study intends to explore the clinicopathological characteristics and survival prognosis of locally recurrent colorectal cancer patients with different treatment modes by retrospectively analyzing the medical records of locally recurrent colorectal cancer patients who received hospitalization in our center. Transcriptome sequencing and public databases were used to screen for molecular markers related to locally recurrent colorectal cancer and to explore molecular markers' regulatory role in the progression of locally recurrent colorectal cancer.

DETAILED DESCRIPTION:
In the past few decades, although the widespread implementation of total mesorectal excision (TME) and neoadjuvant chemoradiotherapy has dramatically reduced the postoperative local recurrence rate of rectal cancer, local recurrence after radical resection of colorectal cancer still affects the long-term survival of patients. One of the main reasons is that the postoperative local recurrence rate in patients with rectal cancer is about 6-10%, while that in colon cancer is about 4-13%. In clinical practice, surgical treatment is the preferred treatment option for patients with locally recurrent colorectal cancer (LRCRC). However, only more than one-third of LRCRC patients can be surgically resected with recurrent lesions. For surgically treatable LRCRC patients, since the recurrent lesions often infiltrate widely, complete resection of the lesions usually requires expanding the scope of surgical resection, and posterior pelvic surgery is needed if necessary. Surgery (PPE) or even total pelvic excision (TPE), the complications, functional impairment, and perioperative death caused by the surgery also affect the patient's near and far prognosis. When there are distant metastases or unresectable recurrent tumors, radical resection is often not feasible, which may result in significant morbidity and mortality, so it is necessary to explore different treatment modalities, especially surgical treatment. What is the impact on LRCRC. The mechanism of local recurrence is usually thought to be caused by insufficient resection margins or the planting of detached tumor cells. Another standard theory is that it is caused by metachronous canceration around the anastomosis.The possible reasons are unstable cell proliferation and epithelial adaptation at the anastomosis site-sexual hyperplasia. Some studies also believe neither theory can explain the higher recurrence rate around the anastomosis, suggesting that it may be due to unique and persistent genetic changes. By reading a large amount of relevant literature, we found that local recurrence is a kind of metastasis or metachronous metastasis. Metastasis is a complex, multi-step process. Current metastasis research mainly focuses on various cancer cells. However, research on the molecular regulatory mechanisms of colorectal cancer metastasis is still limited.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with LRCRC who received hospitalization in our center and patients with stage II-III colorectal cancer whose primary surgery was radical surgery
2. The pathological type of primary tumor is adenocarcinoma
3. Postoperative local recurrence of colorectal cancer diagnosed by imaging or pathological examination
4. Have complete medical records and continuous follow-up records

Exclusion Criteria:

1. Familial hereditary colorectal malignant tumors
2. Past history of other malignant tumors
3. Recurrence and diffuse peritoneal recurrence occurring within 1 month after surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally recurrent colorectal cancer who underwent surgery during hospitalization and whose primary surgical pathology was stage II/III.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3-years
Cancer-specific survival | 3-years

SECONDARY OUTCOMES:
Find a differentially expressed gene | 3-years

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxu Zheng, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Ikoma N, You YN, Bednarski BK, Rodriguez-Bigas MA, Eng C, Das P, Kopetz S, Messick C, Skibber JM, Chang GJ. Impact of Recurrence and Salvage Surgery on Survival After Multidisciplinary Treatment of Rectal Cancer. J Clin Oncol. 2017 Aug 10;35(23):2631-2638. doi: 10.1200/JCO.2016.72.1464. Epub 2017 Jun 28. PMID 28657814
- [Background] Read TE, Mutch MG, Chang BW, McNevin MS, Fleshman JW, Birnbaum EH, Fry RD, Caushaj PF, Kodner IJ. Locoregional recurrence and survival after curative resection of adenocarcinoma of the colon. J Am Coll Surg. 2002 Jul;195(1):33-40. doi: 10.1016/s1072-7515(02)01224-3. PMID 12113543
- [Background] Manfredi S, Bouvier AM, Lepage C, Hatem C, Dancourt V, Faivre J. Incidence and patterns of recurrence after resection for cure of colonic cancer in a well defined population. Br J Surg. 2006 Sep;93(9):1115-22. doi: 10.1002/bjs.5349. PMID 16804870
- [Background] Sjovall A, Granath F, Cedermark B, Glimelius B, Holm T. Loco-regional recurrence from colon cancer: a population-based study. Ann Surg Oncol. 2007 Feb;14(2):432-40. doi: 10.1245/s10434-006-9243-1. Epub 2006 Dec 1. PMID 17139459
- [Background] Yun HR, Lee LJ, Park JH, Cho YK, Cho YB, Lee WY, Kim HC, Chun HK, Yun SH. Local recurrence after curative resection in patients with colon and rectal cancers. Int J Colorectal Dis. 2008 Nov;23(11):1081-7. doi: 10.1007/s00384-008-0530-0. Epub 2008 Aug 8. PMID 18688621
- [Background] Elferink MA, Visser O, Wiggers T, Otter R, Tollenaar RA, Langendijk JA, Siesling S. Prognostic factors for locoregional recurrences in colon cancer. Ann Surg Oncol. 2012 Jul;19(7):2203-11. doi: 10.1245/s10434-011-2183-4. Epub 2012 Jan 5. PMID 22219065
- [Background] Liska D, Stocchi L, Karagkounis G, Elagili F, Dietz DW, Kalady MF, Kessler H, Remzi FH, Church J. Incidence, Patterns, and Predictors of Locoregional Recurrence in Colon Cancer. Ann Surg Oncol. 2017 Apr;24(4):1093-1099. doi: 10.1245/s10434-016-5643-z. Epub 2016 Nov 3. PMID 27812826
- [Background] Pietra N, Sarli L, Thenasseril BJ, Costi R, Sansebastiano G, Peracchia A. Risk factors of local recurrence of colorectal cancer: a multivariate study. Hepatogastroenterology. 1998 Sep-Oct;45(23):1573-8. PMID 9840107
- [Background] Wright HK, Thomas WH, Cleveland JC. The low recurrence rate of colonic carcinoma in ileocolic anastomoses. Surg Gynecol Obstet. 1969 Nov;129(5):960-2. No abstract available. PMID 5824273
- [Background] Phillips RK, Hittinger R, Blesovsky L, Fry JS, Fielding LP. Local recurrence following 'curative' surgery for large bowel cancer: I. The overall picture. Br J Surg. 1984 Jan;71(1):12-6. doi: 10.1002/bjs.1800710104. PMID 6689962
- [Background] Matsuda A, Kishi T, Musso G, Matsutani T, Yokoi K, Wang P, Uchida E. The effect of intraoperative rectal washout on local recurrence after rectal cancer surgery: a meta-analysis. Ann Surg Oncol. 2013 Mar;20(3):856-63. doi: 10.1245/s10434-012-2660-4. Epub 2012 Sep 18. PMID 22987097
- [Result] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Result] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704